CLINICAL TRIAL: NCT02068859
Title: Treatment of Knee Pain With Topical Diclofenac Cream 8% or Diclofenac Gel 1%
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: FPR Specialty Pharmacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FPRSpecialty-0001-CC
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Knee Pain Chronic; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac Cream 8% (Experimental): Diclofenac Cream 8% applied 3-4 times daily for 6 weeks.
  Interventions: Drug: Diclofenac Cream 8%
- Control (Active Comparator): Diclofenac Gel 1% applied 3-4 times daily fr 6 weeks
  Interventions: Drug: Diclofenac Gel 1%

INTERVENTIONS:
Drug: Diclofenac Cream 8% — Subjects will be given instructions to apply the study drug topically 3-4 times daily to the affected knee. Application instructions will also be printed on the tubes of products.
  Arms: Diclofenac Cream 8%
Drug: Diclofenac Gel 1% — Subjects will be given instructions to apply the study drug topically 3-4 times daily to the affected knee. Application instructions will also be printed on the tubes of products.
  Arms: Control

SUMMARY:
Non-steroidal anti-inflammatory medication (NSAID) therapy is a mainstay treatment for joint pain and painful musculoskeletal disorders. Though this form of systemic therapy is highly effective, it causes substantial side effects including gastritis and gastric ulcer disease, renal impairment, hypertension, and thrombotic events. These types of oral medications are utilized by millions of Americans on a fairly regular basis in both over-the-counter preparations and prescription compounds. In recent years, topical preparations of NSAIDs have been used for localized pain as an alternate to oral administration with reported good analgesic efficacy. For example, they are often used for knee pain. There is little systemic absorption of NSAIDs with topical administration, and consequently less likelihood of systemic side effects.

Though much less studied than oral NSAIDs, topical NSAID preparations are currently prescribed for a variety of arthritic and musculoskeletal types of pain. The best-studied commercially available products are diclofenac 1% compounds. Higher concentrations presumably provide higher tissue concentration leading to better and longer pain relief, along with a more prominent anti-inflammatory effect.

The investigators will therefore compare the efficacy of available topical diclofenac 1% gel to that of diclofenac 8% cream. Specifically, the investigators propose to test the hypothesis that efficacy of topical diclofenac 8% exceeds that of diclofenac 1%, without any increase in systemic toxicity.

One hundred six patients presenting to the Cleveland Clinic Pain Management Department for the treatment of knee pain will be randomly assigned to topical diclofenac cream 8% or diclofenac gel 1%, with the designated medication applied the symptomatic area of the knee over 6 weeks. Investigators will be blinded to treatment, and will evaluate pain relief and functional/disability status.

ELIGIBILITY:
Inclusion Criteria:

* Acute and chronic knee pain, along with postoperative knee pain lasting at least two months.

Exclusion Criteria:

* Patients will be excluded if deemed inappropriate for application of topical medication therapy by the treating physician. This will include adult patients with diffuse (non-localized) pain disorders and those likely to need knee surgery during the treatment period.
* Patients with knee infection, open knee wounds, or acute knee skin lesions will be excluded.
* Patients with diclofenac or wheat or gluten allergies will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Descrete Response Scale Pain Scores | Daily measurement for 6 weeks
  Patients will maintain a daily home pain diary. This will be recorded in the evening each day over the six week treatment period with documentation of minimum, maximum, and overall average daily pain on a 0-10/10 discrete response scale (DRS).

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Administration - Outcomes Research, Cleveland, Ohio, United States